CLINICAL TRIAL: NCT04823429
Title: Effects of High Intensity Interval Training and Moderate Intensity Continuous Training on Nitric Oxide-mediated Erythrocyte Rheology
Brief Title: HIIT and MICT on Nitric Oxide-mediated Erythrocyte Rheology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202000448A3
Record Dates: First submitted 2021-02-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Exercise; Interval Training
Keywords: Erythrocyte; eNOS; High intensity interval training; deformability
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity-interval training (HIIT) (Experimental): Subjects performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Interventions: Behavioral: High intensity-interval training (HIIT)
- Moderate intensity-continuous (MICT) (Experimental): Subjects performed MICT (sustained 60%VO 2max) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Interventions: Behavioral: Moderate intensity-continuous (MICT)
- Control group (No Intervention): Without any exercise training

INTERVENTIONS:
Behavioral: High intensity-interval training (HIIT) — Subjects performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Without any exercise training
  Arms: High intensity-interval training (HIIT)
Behavioral: Moderate intensity-continuous (MICT) — Subjects performed MICT (sustained 60%VO 2max) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Arms: Moderate intensity-continuous (MICT)

SUMMARY:
Erythrocyte rheological properties affect blood viscoelasticity and consequently regulate vascular resistance to flow shear force, whereas rheological impairments of erythrocytes may result in circulatory disorders. The aim of this study was to establish an effective exercise strategy for improving individual aerobic capacity and for simultaneously ameliorating the risk of hemorheological dysfunction evoked by a graded exercise test (GXT) and the hypotheses is exercise intervention will improved hemorheological functions by enhancing deformability of erythrocytes via NO-mediated mechanism. This study included 60 healthy sedentary mens (age 20~30) from Chang Gung university than were randomized into the HIIT [3-min intervals at 40% and 80% V̇O2 reserve (V̇O2R),n=10] and MICT(sustained 60% V̇O2R,n=10)on a bicycle ergometer for 30min·d-1, 5 d·wk-1 for 6 wk.

DETAILED DESCRIPTION:
Recently, the role of erythrocyte has been more emphasized, which also related with endothelial cell. For coronary artery patients, the endothelial nitric oxide synthase activity in red blood cell (RBC-eNOS activity) is lower than age-matched health people, and it is related with dysfunction of endothelial cell. In cardiovascular diseases. the erythrocyte arginase-1 is active and seize L-arginine with eNOS. When the Arg-1 stimulated by reactive oxygen species (ROS), the nitric oxide (NO) bioactivity decrease and produce more ROS, meanwhile, ROS can go around to stimulate Arg-1. When the RBC-NO production is lowering, it will increase the adhesion activity to endothelial cell due to erythrocyte can be quite close to blood vessel well then release Nitric Oxide, induce the dysfunction and oxidative pressure of endothelial cell. The NO can also regulate the deformability of erythrocytes, and extremely affect oxygen supply to tissue once the deformability and aggregation of erythrocyte become abnormal. Besides NO, the deformability will be affected if erythrocyte is continuously exposed to the endogenous or exogenous ROS, which also increase adhesion to endothelial cell with the exposure of phosphatidylserine. Exercise can regulate the mechanism of NO release from erythrocyte, affecting the rheology of erythrocyte, and improve the anti-oxidation ability. Therefore, as mentioned above which make erythrocyte, as many aspects, become an important role on atherosclerosis disease treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having a sedentary lifestyle (without regular exercise, exercise frequency ≤ once weekly, duration < 20 min).

Exclusion Criteria:

* Exposed to high altitudes (> 3000 m) for at least 1 year.
* Smoker
* Taking medications or vitamins
* Having any cardiopulmonary/hematological risk.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-09-04 (Estimated); Study Completion 2021-09-04 (Estimated)

PRIMARY OUTCOMES:
Intracellular NO production response to exercise training. | 8 weeks
  Added different inhibitors or agonists to investigate the effects of exercise training on NO production mediated by eNOS-NO pathway.
Intracellular ROS production response to exercise training. | 8 weeks
  Added different inhibitors or agonists to investigate the effects of exercise training on ROS production mediated by eNOS-NO pathway.
The levels of eNOS, p-eNOS and Band-3 response to exercise training. | 8 weeks
  Detect the following protein levels: eNOS, p-eNOS and Band-3, by the western blots.

SECONDARY OUTCOMES:
Determination of erythrocyte biological markers by Flow Cytometry | 8 weeks
  Using the Flow Cytometry to detect the following markers: CD242, CD239, NADPH oxidase 2 (Nox2) and Arginase 1 (Arg1).
Erythrocyte deformability | 8 weeks
  Isolated erythrocyte first, then assess erythrocyte deformability (elongation index ) by using laser assisted optical rotational red cell analyzer (LoRRca).
Cardiopulmonary fitness | 8 weeks
  To assess cardiopulmonary fitness, cardiopulmonary exercise test (CPET) on a cycle ergometer was performed 4 days before and after the intervention. All subjects underwent exercise with a mask to measured oxygen consumption (VO2) breath by breath using a computer-based system.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao TY, Fu LL, Wang JS. Hypoxic exercise training causes erythrocyte senescence and rheological dysfunction by depressed Gardos channel activity. J Appl Physiol (1985). 2011 Aug;111(2):382-91. doi: 10.1152/japplphysiol.00096.2011. Epub 2011 May 5. PMID 21551009
- [Background] Agre P, King LS, Yasui M, Guggino WB, Ottersen OP, Fujiyoshi Y, Engel A, Nielsen S. Aquaporin water channels--from atomic structure to clinical medicine. J Physiol. 2002 Jul 1;542(Pt 1):3-16. doi: 10.1113/jphysiol.2002.020818. PMID 12096044
- [Background] Wang JS, Fu TC, Lien HY, Wang CH, Hsu CC, Wu WC, Chien YW, Cherng WJ. Effect of aerobic interval training on erythrocyte rheological and hemodynamic functions in heart failure patients with anemia. Int J Cardiol. 2013 Sep 30;168(2):1243-50. doi: 10.1016/j.ijcard.2012.11.053. Epub 2012 Nov 27. PMID 23199556
- [Background] Chou SL, Huang YC, Fu TC, Hsu CC, Wang JS. Cycling Exercise Training Alleviates Hypoxia-Impaired Erythrocyte Rheology. Med Sci Sports Exerc. 2016 Jan;48(1):57-65. doi: 10.1249/MSS.0000000000000730. PMID 26672920
- [Background] Grau M, Pauly S, Ali J, Walpurgis K, Thevis M, Bloch W, Suhr F. RBC-NOS-dependent S-nitrosylation of cytoskeletal proteins improves RBC deformability. PLoS One. 2013;8(2):e56759. doi: 10.1371/journal.pone.0056759. Epub 2013 Feb 12. PMID 23424675
- [Background] Suhr F, Brenig J, Muller R, Behrens H, Bloch W, Grau M. Moderate exercise promotes human RBC-NOS activity, NO production and deformability through Akt kinase pathway. PLoS One. 2012;7(9):e45982. doi: 10.1371/journal.pone.0045982. Epub 2012 Sep 25. PMID 23049912